CLINICAL TRIAL: NCT01404559
Title: Metabolic and Biomechanical Measures of Gait Efficiency of Three Multi-Axial, Vertical Shock and Energy Storing-Return Prosthetic Feet During Simple & Complex Mobility Activities
Brief Title: Measures of Gait Efficiency of Three Multi-Axial, Vertical Shock and Energy Storing-Return Prosthetic Feet During Simple & Complex Mobility Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, William Quillen, Associate Dean & Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10193006
Record Dates: First submitted 2011-05-31; First posted 2011-07-28 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Amputation
Keywords: Amputee; Transtibial; Military; Gait; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prosthetic foot 1 (Ossur Variflex) (Active Comparator): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 1 (Ossur Variflex).
  Interventions: Device: Ossur Variflex prosthetic foot
- Prosthetic foot 2 (Ossur Ceterus) (Active Comparator): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 2 (Ossur Ceterus).
  Interventions: Device: Ossur Ceterus prosthetic foot
- Prosthetic foot 3 (Endolite Elite Blade) (Active Comparator): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 3 (Endolite Elite Blade).
  Interventions: Device: Endolite Elite Blade prosthetic foot
- Non-amputee controls (No Intervention): This was an observational arm including non-amputees who were assessed as non-impaired control subjects. There are no interventions in this observational arm of the study.

INTERVENTIONS:
Device: Ossur Variflex prosthetic foot — Lightweight energy-storing prosthetic foot
  Arms: Prosthetic foot 1 (Ossur Variflex)
Device: Ossur Ceterus prosthetic foot — Shock-absorbing prosthetic foot
  Arms: Prosthetic foot 2 (Ossur Ceterus)
Device: Endolite Elite Blade prosthetic foot — Multi-axial prosthetic foot
  Arms: Prosthetic foot 3 (Endolite Elite Blade)

SUMMARY:
Many service members suffering major limb amputation(s) during active duty seek to return to active duty. The purpose of this study is to determine if biomechanic and/or bioenergtic differences exist between popular multi-function prosthetic feet that would facilitate return to duty for soldiers with amputations.

DETAILED DESCRIPTION:
Specific Aims

* Compare the effectiveness of popular prostheses for improving performance in physically demanding tasks and environments.
* Compare amputee performance to a group of high-functioning non-amputees to determine performance differences between the groups.

Hypotheses:

Prosthetic feet with shock absorbing and torsional features will perform better in field activities. Prosthetic feet with high energy return and low mass will perform better during treadmill running. Non-amputee controls will demonstrate superior performance in all outcomes in both field and laboratory environments compared to amputee subjects.

Relevance:

This study has the potential to quantify differences between highly mobile amputees and non-amputees. Additionally, it will provide objective measures of how different prostheses may enhance mobility of soldiers with amputations. The study will compare laboratory and field measures to indicate which conditions increase efficiency of prostheses during rapidly changing mobility demands. This has the potential to permit retention of already trained soldiers.

ELIGIBILITY:
Inclusion Criteria (Amputees):

* Unilateral transtibial amputee ambulating on a K4 prosthesis for >1yr
* K4 functional level
* Currently active duty military or other uniformed service (e.g. police), recently separated Veteran, or strong high-performance athletic history as an amputee (e.g. ranked triathlete, paralympian, etc.)
* Schedule availability and willingness to comply with study protocols
* Aged < 45 years
* Medical clearance, within the last 6 months, for participation in vigorous physical activities

Inclusion Criteria (Non-amputees)

* Currently active duty military, ROTC, or other uniformed service (e.g. police) or recently separated Veteran, or highly accomplished recreational athlete (e.g. marathoner)
* Schedule availability and willingness to comply with study protocols
* Aged < 45 years
* Medical clearance, within the last 6 months, for participation in vigorous physical activities

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Quillen, PT,DPT,PhD, Principal Investigator — University of South Florida; M. Jason Highsmith, PT,DPT,CP, Study Director — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prosthetic Foot 1 (Ossur Variflex): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 1 (Ossur Variflex; 1 week) then prosthetic foot 2(Ossur Ceterus; 1 week) then prosthetic foot 3(Endolite Elite Blade;1 week).
  Ossur Variflex prosthetic foot: Lightweight energy-storing prosthetic foot
- Prosthetic Foot 2 (Ossur Ceterus): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 2(Ossur Ceterus; 1 week) then prosthetic foot 1 (Ossur Variflex; 1 week) then prosthetic foot 3(Endolite Elite Blade; 1 week).
  Ossur Ceterus prosthetic foot: Shock-absorbing prosthetic foot
- Prosthetic Foot 3 (Endolite Elite Blade): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 3(Endolite Elite Blade; 1 week) the prosthetic foot 1(Ossur Variflex; 1 week) then prosthetic foot 2(Ossur Ceterus; 1 week).
  Endolite Elite Blade prosthetic foot: Multi-axial prosthetic foot
- Non-amputee Controls: This was an observational arm including non-amputees who were assessed as non-impaired control subjects. There are no interventions in this observational arm of the study.
  No intervention. Control group.: There are no interventions in this observational arm of the study.
Period: Overall Study
Arm/Group | Prosthetic Foot 1 (Ossur Variflex) | Prosthetic Foot 2 (Ossur Ceterus) | Prosthetic Foot 3 (Endolite Elite Blade) | Non-amputee Controls
Started | 5 | 5 | 4 | 14
Completed | 5 | 5 | 4 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transtibial Amputees: This arm included unilateral transtibial amputees who who were crossed over into 3 different prosthetic feet and assessed per intervention.
- Total: Total of all reporting groups
Arm/Group | Transtibial Amputees | Non-amputee Controls | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.9) | 38.5 (5.1) | 33.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Obstacle Course Completion Time
Description: Laser timing lights were used to measure time necessary to complete a 17 task obstacle course. Participants trigger the laser timing lights when they run past them and the times are recorded in a laptop computer. Laser lights are set up in pairs at the beginning and end of the obstacle course.
Time Frame: 21 days total (7days per prosthetic foot condition)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Prosthetic Foot 1 (Ossur Variflex): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 1.
  Ossur Variflex prosthetic foot: Lightweight energy-storing prosthetic foot
- Prosthetic Foot 2 (Ossur Ceterus): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 2.
  Ossur Ceterus prosthetic foot: Shock-absorbing prosthetic foot
- Prosthetic Foot 3 (Endolite Elite Blade): This arm included unilateral transtibial amputees who who were assessed while using prosthetic foot 3.
  Endolite Elite Blade prosthetic foot: Multi-axial prosthetic foot
Arm/Group | Prosthetic Foot 1 (Ossur Variflex) | Prosthetic Foot 2 (Ossur Ceterus) | Prosthetic Foot 3 (Endolite Elite Blade) | Non-amputee Controls
Number analyzed (Participants) | 14 | 14 | 14 | 14
seconds | 425 (144) | 444 (220) | 419 (130) | 287 (58)

2. Primary Outcome: Bioenergetics Between Feet Components 21 Days After Fitting Prostheses
Description: Measures of energy expenditure while walking on a treadmill were measured. Expired gas (e.g. oxygen and carbon dioxide) are breathed into a face mask worn by participants. The mask contains sensors to detect the levels of the respective gas. Oxygen uptake is correlated with effort to ambulate and therefore, the more oxygen consumed during walking, the more difficult the bout of activity. Thus, if one prosthetic foot requires the consumption of more or less oxygen than other feet, then this is an indicator of the relative difficulty of walking with that particular foot condition.
Time Frame: 21 days total (7days per prosthetic foot condition)
Measure: Mean (Standard Deviation); unit: ml O2/kg/min
Arm/Group | Prosthetic Foot 1 (Ossur Variflex) | Prosthetic Foot 2 (Ossur Ceterus) | Prosthetic Foot 3 (Endolite Elite Blade) | Non-amputee Controls
Number analyzed (Participants) | 14 | 14 | 14 | 14
ml O2/kg/min | 15.7 (2.29) | 15.57 (2.26) | 15.05 (2.17) | 11.05 (1.89)

ADVERSE EVENTS:
Description: Control subjects were not determined to be at risk given that they were not exposed to an intervention and the activities used to measure performance are routine in their daily work and activities.
Groups:
- Unilateral Transtibial Amputees: This arm/group included unilateral transtibial amputees who who were assessed three times. They were exposed to 3 different prosthetic feet interventions.
Arm/Group | Unilateral Transtibial Amputees
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No